CLINICAL TRIAL: NCT02339688
Title: Psychometric Properties of Mobility, Beyond Walking Speed, in Multiple Sclerosis: a Multi-center Study.
Brief Title: Psychometric Properties Mobility Measures MS
Acronym: MCS-III-MOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Dept Neurological Rehabilitation Reha Zentrum Münster Gröben (Unknown); National MS Center Melsbroek (Other); Revalidatie & MS Centrum Overpelt (Other); De Mick (Unknown); Charles University, Czech Republic (Other); Danish MS Hospitals, Haslev and Ry (Other); Masku Neurological Rehabilitation Center (Unknown); Quellenhof (Unknown); Fondazione Don Carlo Gnocchi Onlus (Other); Italian Multiple Sclerosis Foundation (Other); Sheba Medical Center (Other Government); MS-Senteret Hakadal (Unknown); Haukeland University Hospital (Other); MS Rehabilitation Center Borne Sulinowo (Unknown); Clinical center Belgrado (Unknown); Eugenia Epalza Rehabilitation Center, Bilbao, Spain (Other); Cleveland Mellen MS Center (Unknown); University of Colorado, Denver (Other); Queen's University (Other); Shepherd Center Atlanta (Unknown); St. Louis University (Other)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ML10457- S56574
Record Dates: First submitted 2014-12-16; First posted 2015-01-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- convential MS rehabilitation (Other): Investigation of the quality (psychometric properties) and clinical utility of several measures of mobility
  Interventions: Other: conventional MS rehabilitation

INTERVENTIONS:
Other: conventional MS rehabilitation — assessment pre and post conventional MS rehabilitation

SUMMARY:
Current study will investigate the quality (psychometric properties) and clinical utility of several mobility measures, according to disability level. Therefore, several aspects will be inquired:

* Was there an effect of rehabilitation
* Is the measure able to detect change over time? And thus the change exceed measurement error and is it clinically important (responsiveness)
* Does the measure assess what it claims to measure (validity)
* Is the measure able to differentiate all performances of the patients, inclusively the very good and very bad performances (floor and ceiling effects)
* Does the measure gives similar results under consistent test conditions on another testing day (reliability) Worldwide, theoretical approaches to physical therapy and rehabilitation in Multiple Sclerosis often appear significantly different. Since the present research protocol will be performed at different centers across European countries (and US sites), this multi-center study can additionally be applied for mapping the volume and content of rehabilitation, as well as the differential impact of diverse rehabilitation approaches and training volume on mobility, for several disability levels.

Some health-economic analyses will be performed to examine what the approximate cost of rehabilitation compared to effects is and what drivers of costs are (setting, equipment, staff).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to McDonald criteria24,
* Expanded Disability Status Scale25 (EDSS) ≥ 2 and ≤ 6.5 as determined by neurologists or trained clinician
* no relapse within the last month
* no changes in disease modifying treatment and no corticoid-therapy within the last month
* receive at least 10 sessions of physical therapy (in- or outpatient rehabilitation), with a maximum duration of 3 months

Exclusion Criteria:

* other medical conditions interfering with mobility (e.g. stroke, pregnancy, fractures, …)
* other neurological impairments with permanent damage (stroke, Parkinson, …)
* MS-like syndromes such as neuromyelitis optica
* not able to understand and execute simple instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk test (T25FW) | day 1 and at the end of the rehabilitation, an expected average of three months
Timed up and go (TUG), TUGcognitive | day 1 and at the end of the rehabilitation, an expected average of three months
Two minute walk test (2MWT) | day 1 and at the end of the rehabilitation, an expected average of three months
Four Square Step Test (FSST) | day 1 and at the end of the rehabilitation, an expected average of three months
5 repetition sit-to-stand test (5STS-test) | day 1 and at the end of the rehabilitation, an expected average of three months
Modified 5 repetition sit-to-stand test (mod 5STS-test) | day 1 and at the end of the rehabilitation, an expected average of three months
Rivermead Mobility Index (RMI) | day 1 and at the end of the rehabilitation, an expected average of three months
Multiple Sclerosis Walking Scale-12 (MSWS-12) | day 1 and at the end of the rehabilitation, an expected average of three months
Performance Scale mobility (PS-mob) | day 1 and at the end of the rehabilitation, an expected average of three months

SECONDARY OUTCOMES:
Timed Up and Go, manual | day 1 and at the end of the rehabilitation, an expected average of three months
Berg Balance Scale (BBS) | day 1 and at the end of the rehabilitation, an expected average of three months
Dynamic Gait index (DGI) | day 1 and at the end of the rehabilitation, an expected average of three months
Activities-specific Balance Confidence Scale (ABC) | day 1 and at the end of the rehabilitation, an expected average of three months
Trunk Impairment Scale, modified Norwegian version (TIS-modNV) | day 1 and at the end of the rehabilitation, an expected average of three months
International Physical Activity Questionnaire (IPAQ) | day 1 and at the end of the rehabilitation, an expected average of three months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Ilse Baert, Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Belgium